CLINICAL TRIAL: NCT01233128
Title: Association of Vascular Endothelial Growth Factor and LOC387715/HTRA1 Polymorphisms With the Response to Intravitreal Ranibizumab Injections in Polypoidal Choroidal Vasculopathy
Brief Title: Vascular Endothelial Growth Factor (VEGF) & LOC387715/HTRA1 Polymorphism in Polypoidal Choroidal Vasculopathy
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Dong Ho Park, clinical professor, Kyungpook National University Hospital
Other Study IDs: VEGF & LOC387715/HTRA1
Record Dates: First submitted 2010-11-01; First posted 2010-11-03 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2012-04

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Genomic DNA was extracted from peripheral blood with the Qiagen QIAamp Blood Kit (Qiagen, Valencia, CA).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- polypoidal choroidal vasculopathy: patients who were treated for polypoidal choroidal vasculopathy with intravitreal injections of 0.5 mg of ranibizumab monthly for 3 months

SUMMARY:
This study is to investigate whether there is an association of the LOC387715/HTRA1 and vascular endothelial growth factor polymorphism with response to treatment with intravitreal ranibizumab injections for patients with polypoidal choroidal vasculopathy.

DETAILED DESCRIPTION:
This is a retrospective comparative case series comprised of 70 patients being treated for polypoidal choroidal vasculopathy with intravitreal ranibizumab injections and 112 control subjects. Patients were genotyped for the LOC387715 (rs10490924), HTRA1 gene (rs11200638), and VEGF (rs3025039 and rs833069)polymorphism using Real-Time polymerase chain reaction.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 60 years of age at onset
* polyp-like terminal aneurysmal dilations with or without branching vascular networks in ICGA and subretinal reddish-orange protrusions corresponding to polyp-like lesions
* patients who had intravitreal injections of 0.5 mg of ranibizumab monthly for 3 months

Exclusion Criteria:

* patients with retinal or choroidal diseases including pathologic myopia, angioid streaks, idiopathic choroidal neovascularization (CNV), presumed ocular histoplasmosis, and other secondary CNV
* patients who refused genotypic analyses

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The authors did a retrospective chart review of 70 patients with PCV who visited the Department of Ophthalmology, Kyungpook National University Hospital in Daegu, Korea.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2010-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Best-corrected visual acuity | up to 12 months
  Best-corrected visual acuity (BCVA) using the Snellen chart was evaluated including BCVA before treatment and BCVA up to 12 months.

SECONDARY OUTCOMES:
Angiographic characteristics | up to 12 months
  Fluorescein angiography (FA) and ICGA (HRA; Heidelberg Engineering, Dossenheim, Germany)were evaluated. Greatest linear dimension (GLD) was determined based on both FA and ICGA.

CONTACTS AND LOCATIONS:
Overall Officials: In Taek Kim, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- In Taek Kim, Daegu, Kyungsangpookdo, South Korea

REFERENCES:
- [Background] Immonen I, Seitsonen S, Tommila P, Kangas-Kontio T, Kakko S, Savolainen ER, Savolainen MJ, Liinamaa MJ. Vascular endothelial growth factor gene variation and the response to photodynamic therapy in age-related macular degeneration. Ophthalmology. 2010 Jan;117(1):103-8. doi: 10.1016/j.ophtha.2009.06.037. Epub 2009 Nov 6. PMID 19896188
- See also: genetics home reference — http://ghr.nlm.nih.gov/